CLINICAL TRIAL: NCT03276949
Title: Non-Invasive Glucose Measurement Using Raman Spectroscopy During Oral Glucose Tolerance Test
Brief Title: Non-invasive Glucose Measurement Using Laser Technology
Acronym: (Raman)
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Massachusetts Institute of Technology (Other)
Responsible Party: Principal Investigator, Uzma Z Khan, Associate Professor of Medicine, University of Missouri-Columbia
Other Study IDs: 2002948
Record Dates: First submitted 2017-09-05; First posted 2017-09-08 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Oral Glucose Tolerance Test
Keywords: Blood glucose; non-invasive; Raman spectroscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers: Non-diabetic healthy men/women in between age group 18-80 years (all races and ethnicity) will be included for blood glucose measurements
  Interventions: Device: Blood glucose measurement

INTERVENTIONS:
Device: Blood glucose measurement — Device used to measure blood glucose levels
  Other Names: Raman Spectroscopy BLOOD GLUCOSE LEVEL MEASUREMENT

SUMMARY:
This study is to evaluate the capability of Raman spectroscopy as a non-invasive method for monitoring concentrations of glucose by illuminating a small spot on the skin, collecting and analyzing the return light. The glucose measurements obtained by Raman Spectroscopy are correlated with those obtained using YSI glucose analyzer and ACCUCHECK instruments.

DETAILED DESCRIPTION:
Diabetes mellitus (DM), caused by impairment in the glucose metabolism is a worldwide epidemic. It is projected that by the year 2035 there will be approximately 592 million diabetic patients. Blood glucose (BG) levels are finely regulated by insulin secretion and any defects in the secretion or function can lead to DM. As no well-established medical intervention for DM has been known till date, continuous monitoring of BG is the only way to avoid secondary metabolic complications such as strokes, heart attacks, high blood pressure, blindness and coma. Diagnosis and therapeutic monitoring of diabetes requires direct measurement of plasma (or blood) glucose. Measurement of the fasting glucose level is the preferred test for diagnosis of diabetes in children and non-pregnant adults, while the oral glucose tolerance test (OGTT) is the preferred method of diagnosis for gestational diabetes. In addition, patients with an established diagnosis of insulin-dependent diabetes (all type-I and many type-II) require frequent glucose measurements for therapeutic monitoring. Emergence of hand-held glucose sensors have enabled patients with the ability to self-monitor the BG level. The frequent monitoring requires small blood sample (<1 µL) obtained by a "finger-pricking" and electrochemical sensing using a portable 'glucometer'. However the procedure is inconvenient, results in poor patient compliance and lacks in providing real time information about concentration changes. Regardless of the clinical test performed, withdrawal of blood or interstitial fluid is currently required for measurement of BG levels.

The proposed study is based on preliminary research supported by the MIT Laser Biomedical Research Center (LBRC), and promising results obtained with spectroscopic measurement of blood glucose in the laboratory, in an experimental animal model, and in a small cohort of human subject volunteers. In order to make non-invasive glucose measurement a viable clinical technology, however, a methodological implementation and validation from bench to bedside is required. In the application, we propose to accomplish this goal by means of a carefully-designed translational research study employing specifically-designed instrumentation and methods for pre-clinical validation and early clinical studies in human subjects. These studies will incrementally increase in data complexity, culminating in a clinical study in human subjects, as well as a non-invasive, spectroscopic glucose tolerance test as an alternative to OGTT.

ELIGIBILITY:
Inclusion Criteria:

wenty healthy men and women will be studied who will be

* Non diabetic
* Age group between 18 - 80 years
* Prior fasting blood glucose (FBG) values less than or equal to 125 mg/dL
* All races and ethnicity
* Smokers and nonsmokers

Exclusion Criteria:

* Subjects with a known diabetic condition
* With FBG greater than 125 mg/dl or random blood sugar above 200 mg/dL since the study requires observing normal glucose level changes during oral glucose tolerance test.
* Subjects with prior indication of skin irritation or with visible skin rashes
* Any phobia for mechanical device or needle
* Pregnant women will be excluded from the study due to the required blood drawing.
* Children will be excluded as they may not tolerate IV line placement or comply with finger-pricking
* Subjects should not have given blood prior to 8 weeks of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All races and ethnicity
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-04-22 (Actual); Primary Completion 2016-04-29 (Actual); Study Completion 2017-03-13 (Actual)

PRIMARY OUTCOMES:
Non-Invasive Random Glucose Measurement using Raman Spectroscopy during Oral Glucose Tolerance Test | Two weeks
  Blood glucose measurement using Raman spectroscopy

SECONDARY OUTCOMES:
Non-Invasive Random Glucose Measurement using Raman Spectroscopy | Two weeks
  Correlation with Serum and capillary blood glucose measurement

CONTACTS AND LOCATIONS:
Overall Officials: Uzma Khan, MD, Principal Investigator — University of Missouri-Columbia; Anandhi Upendran, Study Director — University of Missouri-Columbia

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with MIT for analysis
Supporting Information: Study Protocol, SAP
Time Frame: One year after publication